CLINICAL TRIAL: NCT05225402
Title: Effects of Norepinephrine on Hemodynamic Measurements of Macrocirculatory and Perfusion Parameters in ICU Patients with Septic Shock
Brief Title: Hemodynamic Measurements of Macrocirculatory and Perfusion Parameters in ICU
Status: Recruiting | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Henrik Wolsted, Doctor, Copenhagen University Hospital, Hvidovre
Other Study IDs: HW-NA-Fluid-Measurements
Record Dates: First submitted 2022-01-12; First posted 2022-02-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock; Hemodynamic Instability; Vasoconstriction
Keywords: Septic Shock; Norepinephrine; Hemodynamic; Microcirculation; Intensive Care
MeSH Terms: conditions — Shock, Septic | interventions — Norepinephrine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Septic Shock: Adult patients with septic shock, admitted to ICUs at Hvidovre and Bispebjerg Hospital, respectively. Sedated and mechanically ventilated adult patients (>18 years).
  Interventions: Drug: Hemodynamic measurements during reduction in Norepinephrine and fluid boli.

INTERVENTIONS:
Drug: Hemodynamic measurements during reduction in Norepinephrine and fluid boli. — 1. Extended monitoring equipment will be connected to the patient. Clinical and biochemical parameters will be collected for a baseline before the next step. A Safety check will be performed to ensure correct patient data, correct equipment function and safety measures are meet. A passive leg raise test will be performed to predict fluid responsiveness, in case of a positive test, a fluid challenge will be administered.
  2. A stepwise reduction of the NE infusion rate from baseline while monitoring stroke volume (SV) to elucidate changes in SV and potential preloadresponsiveness. The reduction will occur in steps of 3-5 minute until either discontinuation of the norepinephrine infusion, a 50% reduction in SV or MAP<40.
  3. While maintaining the NE infusion rate from the previous step 2, a fluid challenge will be administrated, until additional fluid does not increase SV>10%.
  4. As in step 2, a stepwise increase in NE infusion rate to the baseline infusion level or the baseline BP.

SUMMARY:
In septic shock there is growing evidence of a state of hemodynamic "disconnection" with seemingly adequate macrocirculatory values despite actual microcirculation failing to meet cellular demand. Norepinephrine (NE) is recommended as first choice vasoactive agent for the treatment of septic shock. However, the dynamic effects of NE on macro- and microcirculation and perfusion parameters has not been described in detail in the context of septic shock, precluding rational individualized titration of NE and fluids, as recommended recently. In the present prospective observational multicenter study in adult septic shock patients, we intend to explore the effects of NE on preload dependency and tissue perfusion by evaluating the correlation and potential discrepancies between macro- and microcirculation both during titration of NE and after fluid resuscitation. The conclusions drawn from our study will contribute to the physiological knowledge necessary for establishing individualized evidence-based bedside management of hemodynamics in the setting of septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or documented infection
* Need for vasopressors to maintain mean arterial blood pressure (MAP) ≥65 mmHg
* Serum lactate levels >2 mmol/L
* Norepinephrine infusion of > 0.2 mcg/kg/min

Exclusion Criteria:

* Absolute contraindication for esophageal doppler or urinary catheter insertion as noted in the patients' charts.
* Severe valvular pathology and cardiac arrhythmias resulting in severe hemodynamic instability.
* Lithium treatment
* Treatment with other vasopressor or inotropic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 45 adult patients with septic shock according to inclusion criteria admitted to ICUs at Hvidovre and Bispebjerg Hospital, respectively.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Preload responsiveness defined as stroke volume increase > 10%, measured by continuous arterial waveform analysis. | Through study completion, an average of 1 year
  The number of patients who were preload responsive after down-titration of NE.

SECONDARY OUTCOMES:
Cardiac output response measured by lithium indicator dilution and Doppler ultrasound. | Through study completion, an average of 1 year
  The effect on cardiac output after fluid bolus and subsequent up-titration of NE to the pre-intervention blood pressure target.
Microcirculation/perfusion measures during intervention. | Through study completion, an average of 1 year
  The effect of the intervention on measures of tissue perfusion. Different topical sites (Brain, Muscle, Finger, Urethra, Sublingual) by minimal- or noninvasive methods.
CO measurement method | Through study completion, an average of 1 year
  Assess the correlation between indirect measurements of CO and lithium dilution measured CO during NE titration.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No